CLINICAL TRIAL: NCT00274209
Title: Impact of Chromoendoscopy on the Detection of Neoplasia in Ulcerative Colitis
Brief Title: Chromoendoscopy for Ulcerative Colitis Surveillance
Status: Completed | Type: Observational
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Principal Investigator, Michael Chiorean, Associate Professor of Medicine, Indiana University
Organization: Indiana University (Other)
Other Study IDs: 0509-71
Record Dates: First submitted 2006-01-06; First posted 2006-01-10 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Ulcerative Colitis; Crohn's Disease
Keywords: Ulcerative colitis; Crohn's disease; Chromoendoscopy; Dysplasia; Neoplasia
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — endoscopic biopsies
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- IBD patients at risk for neoplasia: Patients with long-standing ulcerative colitis or Crohn's colitis at risk for neoplasia.
  Interventions: Procedure: Chromoendoscopy with magnification

INTERVENTIONS:
Procedure: Chromoendoscopy with magnification — A blue dye (indigo carmine) will be sprayed prior to imaging the bowel lining using a zoom colonoscope. The dye is not absorbed and is safe for human use.

SUMMARY:
Long-standing ulcerative colitis is associated with an increased cancer risk. Chromoendoscopy with dye spraying can detect subtle abnormalities that are not visible with standard endoscopy. The purpose of this study is to determine if chromoendoscopy with fewer "targeted biopsies" can replace standard colonoscopy with multiple "random" biopsies.

DETAILED DESCRIPTION:
Patients with ulcerative colitis (UC) are at increased risk for colon cancer. Current guidelines recommend periodic surveillance colonoscopy in individuals who fulfill certain high-risk criteria. Endoscopists must perform a high number of biopsies (over 33 per patient) in order to increase the yield of such procedures. Chromoendoscopy (CE) has the ability to identify subtle lesions that are otherwise missed by standard endoscopy. Whether CE can replace standard colonoscopy in the surveillance of patients with UC is unknown.

Comparison: both standard biopsies and targeted biopsies will be obtained during colonoscopy from patients with UC who are candidates for surveillance colonoscopy. The yield of the two methods will be compared based on the number of biopsies required to identify one dysplastic (precancerous) lesion.

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative colitis, pancolitis > 8 years; left-sided > 15 years or
* history of PSC or
* history of previous dysplasia on colon biopsies or
* family history of colon cancer in first degree relative

Exclusion Criteria:

* any condition that precludes colonoscopy
* expected survival less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ulcerative colitis satisfying criteria for surveillance colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2005-12; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of dysplastic lesions by white light vs. chromoendoscopy | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael V Chiorean, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Medical Center, Indianapolis, Indiana, United States